CLINICAL TRIAL: NCT03343756
Title: HepaStem Long-Term Safety Registry - Registry for Patients Who Have Been Administered HepaStem
Brief Title: HepaStem Long-Term Safety Registry
Acronym: PROLONGSTEM
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision related to product development prioritisation.
Sponsor: Cellaion SA (Industry)
Responsible Party: Sponsor
Other Study IDs: PROLONGSTEM
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Urea Cycle Disorder; Crigler-Najjar Syndrome; Acute on Chronic Liver Failure
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Crigler-Najjar Syndrome; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients having received at least one infusion of the Investigational Medicinal Product (IMP) HepaStem HHALPC during a previous interventional clinical study conducted by Promethera Biosciences

ELIGIBILITY:
Inclusion Criteria:

* All patients having received at least one infusion of HepaStem during a previous interventional clinical study conducted by Promethera.

Exclusion Criteria:

* Patients who received an OLT and completed 6-month FU documentation prior to the start of the PROLONGSTEM study.
* Patients who have received mature liver cells or stem cells other than HepaStem prior to the start of the PROLONGSTEM study.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received HepaStem in the interventional studies conducted by Promethera will be proposed to participate in this PROLONGSTEM study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events of Specific Interest (AESI) | 60 months
  Adverse Events of Specific Interest (AESI):
  * Event with fatal outcome (Death)
  * Orthotopic Liver Transplantation (OLT) and Outcome.
  * Development of Malignancy or unwanted tissue formation in different organs (tumor malignant or not).
  * Disease linked to transmission of adventitious agents or reactivation of latent pathogens.
  * Any AE which in the opinion of the Investigator has a plausible causal relationship to HepaStem.

CONTACTS AND LOCATIONS:
Locations (29):
- Belgium (8):
  - Hopital Erasme, Anderlecht
  - Antwerp University Hospital, Antwerp
  - Association Hospitaliere De Bruxelles Et De Schaerbeek Centre Hospitalier Universitaire Brugmann, Brussels
  - UCL, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHC MontLegia, Liège
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Bulgaria (3):
  - University Multiprofile Hospital For Active Treatment Dr. Georgi Stranski EAD, Pleven
  - UMHAT Medica Ruse, Rousse
  - Military Medical Academy, Sofia
- France (11):
  - Centre Hospitalier Universitaire Amiens Picardie, Amiens
  - Centre Hospitalier Universitaire D'Angers, Angers
  - University Hospital Of Bordeaux, Bordeaux
  - CHU Lille, Lille
  - Hospices Civils De Lyon, Lyon
  - Assistance Publique Hopitaux De Marseille, Marseille
  - Centre Hospitalier Universitaire De Montpellier, Montpellier
  - Assistance Publique Hopitaux De Paris, Paris
  - Les Hopitaux Universitaires De Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - Hopital Paul Brousse, Villejuif
- Id Clinic, Mysłowice, Poland
- Spain (6):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Parc Tauli Hospital Universitari, Sabadell
  - Hospital Unviersitario Miguel Servet, Zaragoza